CLINICAL TRIAL: NCT06195475
Title: Impact of Tidal Volume Magnitude in Pressure Support Mode on Mortality in Adults Under Invasive Mechanical Ventilation. Multi-center Retrospective Cohort Study.
Brief Title: Association Between Tidal Volume and Mortality in Pressure Support in Adults Under Invasive Mechanical Ventilation
Acronym: SAFE-VT
Status: Completed | Type: Observational
Sponsor: Sanatorio Anchorena San Martin (Other)
Collaborators: Javier Hernán Dorado (Unknown); Joaquin Perez (Unknown)
Responsible Party: Principal Investigator, Matias Accoce, Respiratory and physical therapist, Sanatorio Anchorena San Martin
Other Study IDs: Sanatorio Anchorena San Martín
Record Dates: First submitted 2023-10-03; First posted 2024-01-08 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Respiration, Artificial
Keywords: pressure support ventilation; tidal volume
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- exposure to tidal volumes greater than 8 ml/kg of predicted body weight: exposure to tidal volumes greater than 8 ml/kg of predicted body weight during the initial 48 hours of pressure support mode mechanical ventilation
  Interventions: Other: high vs low tidal volume
- tidal volume equal to or less than 8 ml/kg of predicted body weight: individuals who maintain a tidal volume equal to or less than 8 ml/kg of predicted body weight
  Interventions: Other: high vs low tidal volume

INTERVENTIONS:
Other: high vs low tidal volume — The clinical investigation aims to determine whether exposure to tidal volumes greater than 8 ml/kg of predicted body weight during the initial 72 hours of pressure support mode mechanical ventilation is associated with an increased risk of mortality in the intensive care unit when compared to individuals who maintain a tidal volume equal to or less than 8 ml/kg of predicted body weight.

SUMMARY:
The goal of this Multicenter retrospective cohort study is to assessing the association between the development of a tidal volume magnitude > 8 ml/kg of predicted body weight during the first transition to partial support phase in pressure support mode and mortality in the intensive care unit in a general population of patients older than 18 years who require invasive mechanical ventilation, in contrast to individuals who develop tidal volume ≤ 8 ml/kg of predicted body weight. Secondarily, assess the association between elevated VT (tidal volume) during the initiation of the partial support phase in pressure support mode and ventilator-free days, failure in transitioning to spontaneous ventilation, and success in weaning from mechanical ventilation.

The main question it aims to answer are:

• Does exposure to tidal volumes greater than 8 ml/kg of predicted body weight during the first 48 hours of pressure support mode mechanical ventilation increase the risk of death in the intensive care unit compared to those who develop a tidal volume equal to or less than 8 ml/kg of predicted body weight in subjects older than 18 years requiring invasive mechanical ventilation?

The clinical investigation aims to determine whether exposure to tidal volumes greater than 8 ml/kg of predicted body weight during the initial 48 hours of pressure support mode mechanical ventilation is associated with an increased risk of mortality in the intensive care unit when compared to individuals who maintain a tidal volume equal to or less than 8 ml/kg of predicted body weight. This analysis involves subjects aged 18 years and older who require invasive mechanical ventilation

DETAILED DESCRIPTION:
The data of patients from each participating center in the study will be encoded to maintain their anonymity. These center-related data will only be known to the study's Principal Investigator (PI), who will be the sole individual with access to them. Under no circumstances will the centers be able to make comparisons among themselves.

The data collected by each participating unit will be gathered by the investigator or by one of the designated team members assigned to the study, and entered into a REDCap® form specifically designed for this study.

The data collected by each investigator will be randomly supervised by the coordinating group to ensure the quality of the collected data and to detect possible errors in data acquisition. The study's coordinating group will also monitor the daily incorporation of data into the database to supervise and detect, as a double filter, the possibility of errors in data editing and incorporation, thus ensuring the quality and reliability of the information obtained throughout the entire period of patient inclusion.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 and older admitted to the participating ICUs from January 1, 2019, to April 30, 2023, with a requirement for mechanical ventilation (MV) for any reason for at least 72 hours within the same cycle, who have at least one monitoring session in PC-CSV (pressure support ventilation), and who remain on MV (regardless of the mode) for a period of ≥ 1 calendar day after that monitoring session will be included

Exclusion Criteria:

* Patients who have not initiated the partial support phase in PC-CSV mode or who are extubated within a period of less than 24 hours from the first ventilatory monitoring in PC-CSV will be excluded. Subjects with missing data in exposure and/or outcome variables will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years or older in invasive mechanical ventilation who have remained in PC-CSV for at least 24 hours
Sampling Method: Non-Probability Sample
Enrollment: 2607 (Actual)
Dates: Start 2023-11-30 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
mortality in intensive care unit | day 28
  Categorical dichotomous variable (yes/no). All patients who are discharged from the intensive care unit (ICU), regardless of their destination (another area within the institution or another healthcare facility of any kind), will be considered as alive at ICU discharge.

SECONDARY OUTCOMES:
Failure in transitioning to spontaneous ventilation | 72 hours
  Categorical dichotomous variable (yes/no). It will be considered a failure in transitioning to spontaneous ventilation for any subject who, after having at least one monitoring session in PC-CSV mode, has at least one monitoring session in mandatory modes (VC-CMV and/or PC-CMV) within the following 72 hours.
Ventilator-free days | 28 days
  Discrete quantitative variable. To count each day of mechanical ventilation (MV), daily programming and respiratory mechanics monitoring will be used; considering one monitoring session as one day of MV. To obtain the final variable, the following equation will be used: 28 - days of invasive MV, resulting in a possible data range from 0 to 26 ventilator-free days.
ICU length of stay | 28 days
  Discrete quantitative variable. It will be obtained using the following equation: (Date of ICU discharge) - (Date of ICU admission). Only the number of days of hospitalization will be required for the analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Sanatorio Anchorena San Martín, Buenos Aires, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Litell JM, Gong MN, Talmor D, Gajic O. Acute lung injury: prevention may be the best medicine. Respir Care. 2011 Oct;56(10):1546-54. doi: 10.4187/respcare.01361. PMID 22008396
- [Background] Acute Respiratory Distress Syndrome Network; Brower RG, Matthay MA, Morris A, Schoenfeld D, Thompson BT, Wheeler A. Ventilation with lower tidal volumes as compared with traditional tidal volumes for acute lung injury and the acute respiratory distress syndrome. N Engl J Med. 2000 May 4;342(18):1301-8. doi: 10.1056/NEJM200005043421801. PMID 10793162
- [Background] Gajic O, Dara SI, Mendez JL, Adesanya AO, Festic E, Caples SM, Rana R, St Sauver JL, Lymp JF, Afessa B, Hubmayr RD. Ventilator-associated lung injury in patients without acute lung injury at the onset of mechanical ventilation. Crit Care Med. 2004 Sep;32(9):1817-24. doi: 10.1097/01.ccm.0000133019.52531.30. PMID 15343007
- [Background] Serpa Neto A, Cardoso SO, Manetta JA, Pereira VG, Esposito DC, Pasqualucci Mde O, Damasceno MC, Schultz MJ. Association between use of lung-protective ventilation with lower tidal volumes and clinical outcomes among patients without acute respiratory distress syndrome: a meta-analysis. JAMA. 2012 Oct 24;308(16):1651-9. doi: 10.1001/jama.2012.13730. PMID 23093163
- [Background] Hubmayr RD, Kallet RH. Understanding Pulmonary Stress-Strain Relationships in Severe ARDS and Its Implications for Designing a Safer Approach to Setting the Ventilator. Respir Care. 2018 Feb;63(2):219-226. doi: 10.4187/respcare.05900. PMID 29367383
- [Background] Murias G, Lucangelo U, Blanch L. Patient-ventilator asynchrony. Curr Opin Crit Care. 2016 Feb;22(1):53-9. doi: 10.1097/MCC.0000000000000270. PMID 26627539
- [Background] Plotnikow GA, Gogniat E, Accoce M, Navarro E, Dorado JH; EpVAr study group. Epidemiology of mechanical ventilation in Argentina. The EpVAr multicenter observational study. Med Intensiva (Engl Ed). 2022 Jul;46(7):372-382. doi: 10.1016/j.medine.2022.05.002. Epub 2022 May 31. PMID 35660286
- [Background] Kress JP, Pohlman AS, O'Connor MF, Hall JB. Daily interruption of sedative infusions in critically ill patients undergoing mechanical ventilation. N Engl J Med. 2000 May 18;342(20):1471-7. doi: 10.1056/NEJM200005183422002. PMID 10816184
- [Background] Girard TD, Kress JP, Fuchs BD, Thomason JW, Schweickert WD, Pun BT, Taichman DB, Dunn JG, Pohlman AS, Kinniry PA, Jackson JC, Canonico AE, Light RW, Shintani AK, Thompson JL, Gordon SM, Hall JB, Dittus RS, Bernard GR, Ely EW. Efficacy and safety of a paired sedation and ventilator weaning protocol for mechanically ventilated patients in intensive care (Awakening and Breathing Controlled trial): a randomised controlled trial. Lancet. 2008 Jan 12;371(9607):126-34. doi: 10.1016/S0140-6736(08)60105-1. PMID 18191684
- [Background] van Haren F, Pham T, Brochard L, Bellani G, Laffey J, Dres M, Fan E, Goligher EC, Heunks L, Lynch J, Wrigge H, McAuley D; Large observational study to UNderstand the Global impact of Severe Acute respiratory FailurE (LUNG SAFE) Investigators. Spontaneous Breathing in Early Acute Respiratory Distress Syndrome: Insights From the Large Observational Study to UNderstand the Global Impact of Severe Acute Respiratory FailurE Study. Crit Care Med. 2019 Feb;47(2):229-238. doi: 10.1097/CCM.0000000000003519. PMID 30379668
- [Background] Pinto EF, Santos RS, Antunes MA, Maia LA, Padilha GA, de A Machado J, Carvalho ACF, Fernandes MVS, Capelozzi VL, de Abreu MG, Pelosi P, Rocco PRM, Silva PL. Static and Dynamic Transpulmonary Driving Pressures Affect Lung and Diaphragm Injury during Pressure-controlled versus Pressure-support Ventilation in Experimental Mild Lung Injury in Rats. Anesthesiology. 2020 Feb;132(2):307-320. doi: 10.1097/ALN.0000000000003060. PMID 31939846
- [Background] Henzler D, Schmidt A, Xu Z, Ismaiel N, Zhang H, Slutsky AS, Pelosi P. Increased effort during partial ventilatory support is not associated with lung damage in experimental acute lung injury. Intensive Care Med Exp. 2019 Nov 5;7(1):60. doi: 10.1186/s40635-019-0272-z. PMID 31691042
- [Background] Perez J, Dorado JH, Papazian AC, Berastegui M, Gilgado DI, Cardoso GP, Cesio C, Accoce M. Titration and characteristics of pressure-support ventilation use in Argentina: an online cross-sectional survey study. Rev Bras Ter Intensiva. 2020 Mar;32(1):81-91. doi: 10.5935/0103-507x.20200013. Epub 2020 May 8. PMID 32401994
- [Background] Bellani G, Grassi A, Sosio S, Gatti S, Kavanagh BP, Pesenti A, Foti G. Driving Pressure Is Associated with Outcome during Assisted Ventilation in Acute Respiratory Distress Syndrome. Anesthesiology. 2019 Sep;131(3):594-604. doi: 10.1097/ALN.0000000000002846. PMID 31335543
- [Background] Yoshida T, Fujino Y, Amato MB, Kavanagh BP. Fifty Years of Research in ARDS. Spontaneous Breathing during Mechanical Ventilation. Risks, Mechanisms, and Management. Am J Respir Crit Care Med. 2017 Apr 15;195(8):985-992. doi: 10.1164/rccm.201604-0748CP. PMID 27786562
- [Background] Esteban A, Frutos-Vivar F, Muriel A, Ferguson ND, Penuelas O, Abraira V, Raymondos K, Rios F, Nin N, Apezteguia C, Violi DA, Thille AW, Brochard L, Gonzalez M, Villagomez AJ, Hurtado J, Davies AR, Du B, Maggiore SM, Pelosi P, Soto L, Tomicic V, D'Empaire G, Matamis D, Abroug F, Moreno RP, Soares MA, Arabi Y, Sandi F, Jibaja M, Amin P, Koh Y, Kuiper MA, Bulow HH, Zeggwagh AA, Anzueto A. Evolution of mortality over time in patients receiving mechanical ventilation. Am J Respir Crit Care Med. 2013 Jul 15;188(2):220-30. doi: 10.1164/rccm.201212-2169OC. PMID 23631814
- [Background] Abrams D, Montesi SB, Moore SKL, Manson DK, Klipper KM, Case MA, Brodie D, Beitler JR. Powering Bias and Clinically Important Treatment Effects in Randomized Trials of Critical Illness. Crit Care Med. 2020 Dec;48(12):1710-1719. doi: 10.1097/CCM.0000000000004568. PMID 33031148
- See also: Mark Stevenson, Evan Sergeant with contributions from Telmo Nunes, Cord Heuer, Jonathon Marshall, Javier Sanchez, Ron Thornton, Jeno Reiczigel, Jim Robison-Cox, Paola Sebastiani, Peter Solymos, Kazuki Yoshida, Geoff Jones, Sarah Pirika — https://CRAN.R-project.org/package=epiR